CLINICAL TRIAL: NCT02024087
Title: A Phase 1b, Open Label Study of Dalantercept Plus Sorafenib in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Study of Dalantercept and Sorafenib in Patients With Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A041-05; ACE-041
Record Dates: First submitted 2013-12-20; First posted 2013-12-31 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2021-02

CONDITIONS: Advanced Adult Hepatocellular Carcinoma
MeSH Terms: interventions — ALK1-Fc fusion protein, human; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dalantercept 0.6 mg/kg plus sorafenib 400 mg (Experimental): Cohort 1: Participants received dalantercept 0.6 mg/kg by subcutaneous (SC) injection once every 3 weeks plus sorafenib 400 mg orally (PO) once daily
  Interventions: Drug: Dalantercept plus sorafenib
- Dalantercept 0.4 mg/kg plus sorafenib 400 mg (Experimental): Cohort 2: Participants will receive dalantercept 0.4 mg/kg SC injection once every 3 weeks plus sorafenib 400 mg PO once daily
  Interventions: Drug: Dalantercept plus sorafenib
- Expansion cohort - dalantercept 0.4 mg/kg plus sorafenib 400 mg (Experimental): Cohort 3: Participants will receive dalantercept 0.4 mg/kg SC injection once every 3 weeks plus sorafenib 400 mg PO once daily
  Interventions: Drug: Dalantercept plus sorafenib

INTERVENTIONS:
Drug: Dalantercept plus sorafenib — Subcutaneous (SC) injection of dalantercept once every 3 weeks and oral sorafenib daily.
  Other Names: ACE-041

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of dalantercept plus sorafenib in patients with advanced hepatocellular carcinoma (HCC) to determine the recommended dose level of dalantercept in combination with sorafenib.

DETAILED DESCRIPTION:
The initial design of the study was a dose escalating approach in which dalantercept in combination with sorafenib, would be administered at increasing dose levels among 3 cohorts of subjects with HCC in order to determine the Maximum Tolerated Dose (MTD) of the combination. Once the MTD was determined, a forth expansion cohort of subjects would be enrolled at the MTD to assess safety. A total of up to 38 subjects were planned.

The initial cohort (Cohort 1) enrolled 5 subjects at a dalantercept dose level of 0.6 mg/kg once every 3 weeks (Q3W) in combination with sorafenib (400 mg PO once daily). Following an assessment of safety/tolerability by a Safety Review Team, it was recommended to de-escalate the dalantercept dose for Cohort 2 to 0.4 mg/kg Q3W in combination with sorafenib (400 mg PO once daily); 6 subjects were enrolled.

The 0.4 mg/kg dose level was determined to be the MTD, and an additional 10 subjects were enrolled at that dose level in the expansion cohort (Cohort 3).

A formal Statistical Analysis Plan was initially planned for this study. However, due to its early termination, only cursory descriptive statistics were carried out on the available data; no formal SAP was prepared.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, locally advanced or metastatic HCC.
* Child-Pugh Score A (5-6)
* At least one target lesion that has not been treated with local therapy and is measurable by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Life expectancy of at least 12 weeks.
* Able to tolerate oral therapy.
* Appropriate clinical laboratory values within 72 hours prior to study day 1:
* Females of child bearing potential (defined as sexually mature women who have not undergone hysterectomy or bilateral oophorectomy, or are not naturally postmenopausal ≥ 24 consecutive months) must have negative urine or blood pregnancy test prior to enrollment and use adequate birth control methods (abstinence, oral contraceptives, barrier method with spermicide, or surgical sterilization) during study participation. Males must agree to use a latex condom during any sexual contact with females of child bearing potential while participating in the study and for 12 weeks following the last dose of dalantercept, even if he has undergone a successful vasectomy. Patients must be counseled concerning measures to be used to prevent pregnancy and potential toxicities prior to the first dose of dalantercept.

Exclusion Criteria:

* Mixed tumor histology
* Prior systemic therapy for metastatic disease.
* Adjuvant therapy < 6 months prior to study day 1.
* Prior treatment with dalantercept or other agent targeting the ALK1 pathway.
* Prior treatment with sorafenib or other RAF/VEGF targeted therapies.
* Hepatic radiation, chemoembolization, and radiofrequency ablation < 4 weeks prior to study day 1.
* Palliative radiation therapy to metastatic sites of disease < 2 weeks prior to study day 1.
* Interferon therapy < 4 weeks prior to study day 1.
* Uncontrolled Hepatitis B despite appropriate therapy.
* Clinically significant pulmonary, endocrine, neurologic, hematologic, gastrointestinal (GI), autoimmune, psychiatric or genitourinary disease unrelated to HCC that in the judgment of the investigator should preclude treatment with dalantercept or sorafenib.
* Known HIV infection.
* Clinically significant cardiovascular risk
* Clinically significant active pulmonary risk
* Known active gastrointestinal (GI) bleeding.
* Known bleeding diathesis Known history of hereditary hemorrhagic telangiectasia (HHT).
* History of another primary cancer, with the exception of:

  1. Curatively resected non melanoma skin cancer.
  2. Curatively treated cervical carcinoma in situ.
  3. Other primary solid tumor with no known active disease in the opinion of the investigator that will not affect patient outcome in the setting of current HCC diagnosis.
* Major surgery within 4 weeks prior to study day 1 Active infection Anti-coagulation therapy Concomitant treatment with potent CYP3A4 inducers
* Peripheral edema ≥ grade 2 within 2 weeks prior to study day 1.
* History of recurrent ascites requiring paracentesis within 4 weeks of study day 1.
* History of severe (using the National Cancer Institute Common Toxicity Criteria for Adverse Events, version 4.0 [NCI-CTCAE] v4 current minor version ≥ grade 3) allergic or anaphylactic reaction or hypersensitivity to recombinant proteins or excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-08-04 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-09-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Kansas Medical Center (KUMC), Westwood, Kansas
  - Beth Israel Deaconess Medical Center (BIDMC), Boston, Massachusetts
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio

REFERENCES:
- [Derived] Abou-Alfa GK, Miksad RA, Tejani MA, Williamson S, Gutierrez ME, Olowokure OO, Sharma MR, El Dika I, Sherman ML, Pandya SS. A Phase Ib, Open-Label Study of Dalantercept, an Activin Receptor-Like Kinase 1 Ligand Trap, plus Sorafenib in Advanced Hepatocellular Carcinoma. Oncologist. 2019 Feb;24(2):161-e70. doi: 10.1634/theoncologist.2018-0654. Epub 2018 Oct 23. PMID 30352941

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled 04-AUG-2014 Last subject completed 05-JUL-2017 Study conducted at academic oncology centers in the US
Groups:
- Dalantercept 0.6 mg/kg Plus Sorafenib 400 mg: Cohort 1: Participants were administered dalantercept 0.6 mg/kg by subcutaneous injection once every 3 weeks and sorafenib 400 mg orally once daily
- Dalantercept 0.4 mg/kg Plus Sorafenib 400 mg: Cohort 2: Participants were administered dalantercept 0.4 mg/kg by subcutaneous injection once every 3 weeks and sorafenib 400 mg orally once daily
Period: Overall Study
Arm/Group | Dalantercept 0.6 mg/kg Plus Sorafenib 400 mg | Dalantercept 0.4 mg/kg Plus Sorafenib 400 mg
Started | 5 | 16 (Dose change to 0.4 mg/kg and cohort expanded to 16 participants in total at this dose level)
Completed | 5 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dalantercept 0.6 mg/kg Plus Sorafenib 400 mg: Cohort 1: participants were administered dalantercept 0.6 mg/kg by subcutaneous injection once every 3 weeks plus sorafenib 400 mg orally once daily
- Dalantercept 0.4 mg/kg Plus Sorafenib 400 mg: Cohort 2: participants were administered dalantercept 0.4 mg/kg by subcutaneous injection once every 3 weeks plus sorafenib 400 mg orally once daily
- Total: Total of all reporting groups
Arm/Group | Dalantercept 0.6 mg/kg Plus Sorafenib 400 mg | Dalantercept 0.4 mg/kg Plus Sorafenib 400 mg | Total
Number analyzed (Participants) | 5 | 16 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 9 | 11
  >=65 years | 3 | 7 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (16.9) | 64.3 (10.1) | 64.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 3 | 11 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 2 | 15 | 17
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 16 | 21
ECOG status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) status is used by healthcare professionals to assess how a patient's disease is progressing, assess how the disease affects the daily living abilities of the patient, and determine appropriate treatment and prognosis.
  A score of 0 indicates that a participant is fully active, able to carry on all pre-disease performance without restriction.
  A score of 1 indicate that a participant is restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    ECOG 1 | 4 | 8 | 12
    ECOG 0 | 1 | 8 | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events as a Measure of Safety and Tolerability.
Description: Assessed by monitoring AEs using the current active minor version on the National Cancer Institute Common Toxicity Criteria for Adverse Events, version 4.0 (NCI-CTCAE v4 current minor version), physical examinations, vital signs, clinical laboratory test, ECHO, ECG and ADA testing; through final study visit, up to approximately 20 weeks from first dose of dalantercept.
Time Frame: up to approximately 20 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Dalantercept 0.4 mg/kg Plus Sorafenib; Dalantercept 0.6 mg/kg Plus Sorafenib: Dalantercept plus sorafenib: Subcutaneous (SC) injection of dalantercept once every 3 weeks and oral sorafenib daily.
Arm/Group | Dalantercept 0.4 mg/kg Plus Sorafenib | Dalantercept 0.6 mg/kg Plus Sorafenib
Number analyzed (Participants) | 16 | 5
Participants | 16 | 5

2. Secondary Outcome: Best Overall Response
Description: The Best Overall Response (BOR) is the best response recorded from the start of the study treatment until the disease progression/recurrence, scored as one of the following: Complete Response (CR); Partial Response (PR); Stable Disease (SD) or Progressive Disease (PD).
  Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.1), a CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. A PR is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study. PD is defined as At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study.
Time Frame: up to approximately 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dalantercept 0.4 mg/kg Plus Sorafenib | Dalantercept 0.6 mg/kg Plus Sorafenib
Number analyzed (Participants) | 15 | 3
Participants
  Complete response | 0 | 0
  Partial response | 0 | 0
  Stable disease | 8 | 2
  Progressive disease | 7 | 1

3. Secondary Outcome: Overall Survival (OS)
Description: The proportion of participants alive from the initiation of treatment through end of study
Time Frame: up to approximately 20 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Dalantercept 0.6 mg/kg Plus Sorafenib: Dalantercept plus sorafenib: Subcutaneous (SC) injection of dalantercept once every 3 weeks
Arm/Group | Dalantercept 0.4 mg/kg Plus Sorafenib | Dalantercept 0.6 mg/kg Plus Sorafenib
Number analyzed (Participants) | 16 | 5
Participants | 7 | 0

4. Secondary Outcome: Disease Control Rate (DCR)
Description: Percentage of patients whose disease improves or remains stable over a certain time period. DCR is the sum of the complete, partial and stable disease rates.
Time Frame: up to approximately 20 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dalantercept 0.4 mg/kg Plus Sorafenib | Dalantercept 0.6 mg/kg Plus Sorafenib
Number analyzed (Participants) | 15 | 3
Participants | 8 | 2

ADVERSE EVENTS:
Time Frame: Adverse event data were collection from the date of first patient enrollment to the end-of study visit (approximately 20 weeks)
Arm/Group | Dalantercept 0.4 mg/kg Plus Sorafenib | Dalantercept 0.6 mg/kg Plus Sorafenib
All-Cause Mortality (participants affected / at risk) | 9/16 | 5/5
Serious Adverse Events (participants affected / at risk) | 6/16 | 4/5
Other Adverse Events (participants affected / at risk) | 16/16 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalantercept 0.4 mg/kg Plus Sorafenib (N=16) | Dalantercept 0.6 mg/kg Plus Sorafenib (N=5)
abdominal pain (Gastrointestinal disorders) | 2 | 2
atrial fibrillation (Cardiac disorders) | 1 | 1
haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
ejection fraction decrease (Investigations) | 0 | 1
hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dalantercept 0.4 mg/kg Plus Sorafenib (N=16) | Dalantercept 0.6 mg/kg Plus Sorafenib (N=5)
abdominal pain (Gastrointestinal disorders) | 6 | 1
peripheral oedema (General disorders) | 4 | 2
pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
leukopoenia (Blood and lymphatic system disorders) | 3 | 1
asthenia (General disorders) | 2 | 0
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-04): https://cdn.clinicaltrials.gov/large-docs/87/NCT02024087/Prot_SAP_001.pdf